CLINICAL TRIAL: NCT04120376
Title: An Emergency Department-Based Study to Reduce Adolescent Pregnancy
Brief Title: Reducing Adolescent Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other); University of Pittsburgh (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-016314; 5R21HD095096-02 (NIH)
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy in Adolescence; Counseling; Contraception Behavior
Keywords: Contraception counseling; Adolescent pregnancy; Contraception initiation
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Contraception counseling will occur for all adolescent participants and APPs will be enrolled to conduct counseling. The number of participants enrolled includes the final number of participants including adolescent and APPs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counseling Intervention (Experimental): All participants will receive contraception counseling by study Advanced Practice Providers (APPs)
  Interventions: Behavioral: Contraception Counseling

INTERVENTIONS:
Behavioral: Contraception Counseling — Each participant will receive a 10 minute confidential contraception counseling session with an APP in the Emergency Department

SUMMARY:
This multi-site study is employing a brief contraception counseling intervention in the Emergency Department (ED) to shed light on factors that affect decision making as well as barriers and facilitators to conception initiation in the Emergency Department (ED) setting. The overarching goal of the study is to reduce unintended pregnancy among females ages 15 to 18 who present to the Emergency Department (ED).

DETAILED DESCRIPTION:
This study is a prospective cohort study involving females who present to one of two emergency departments (ED) between the ages of 16 and 18, who are at risk of unintended pregnancy.

Our primary objective is to assess intention to initiate contraception ("high"=very/somewhat likely vs "low"=unsure/not likely/definitely not on Likert scale survey) among females aged 15 to 18 years who receive emergency department-based contraceptive counseling.

Our secondary objectives are as follows:

1. Among the same population, assess completion of a referral for any contraceptive care, defined as attendance at a referral site within 4 weeks after the index ED visit.
2. Assess the proportion who ultimately initiate contraception through electronic medical record documentation (i.e., visit note, procedure note, medication review) and participant report (follow-up calls).
3. Use qualitative interview methodology to explore attitudes, barriers, and facilitators that affect decisions to A) express intention to initiate contraception, B) complete a referral for contraceptive care, and C) ultimately initiate contraception among this unique group of high-risk adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 15-18 years who are at high-risk of pregnancy, defined as sexual activity within the last 6 months or likely future sexual activity.
2. Females who do not desire to become pregnant within the next year.
3. Eligible individuals must be proficient in speaking and reading in English.
4. Consent of the adolescent.

Exclusion Criteria:

1. Females who are currently using hormonal contraception or an intrauterine device.
2. Females who are pregnant.
3. Patient has a developmental delay limiting participation.
4. Patient is presenting in the ED after sexual assault.
5. Patient is too ill to be screened.

APPs: [no age limit]] Have been working in ED 6 months

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Individuals who identify as females and are at risk of getting pregnant.
Enrollment: 144 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Mollen, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Only the site PIs and team will have access to study data.

REFERENCES:
- [Background] Hoffman SD, Maynard RA. Kids having kids: Economic costs & social consequences of teen pregnancy. The Urban Institute; 2008.
- [Background] Teen Childbearing Cost Taxpayers $9.4 Billion in 2010 [press release]. 2013.
- [Background] Miller E, Goldstein S, McCauley HL, Jones KA, Dick RN, Jetton J, Silverman JG, Blackburn S, Monasterio E, James L, Tancredi DJ. A school health center intervention for abusive adolescent relationships: a cluster RCT. Pediatrics. 2015 Jan;135(1):76-85. doi: 10.1542/peds.2014-2471. Epub 2014 Dec 22. PMID 25535265
- [Background] Guttmacher Institute. Adolescent pregnancy and its outcomes across countries. Fact Sheet; August 2015. https://www.guttmacher.org/fact-sheet/adolescent-pregnancy-and-its-outcomes-across-countries; accessed January 12, 2018.
- [Background] Lindberg L, Santelli J, Desai S. Understanding the Decline in Adolescent Fertility in the United States, 2007-2012. J Adolesc Health. 2016 Nov;59(5):577-583. doi: 10.1016/j.jadohealth.2016.06.024. Epub 2016 Aug 29. PMID 27595471
- [Background] Santelli JS, Lindberg LD, Finer LB, Singh S. Explaining recent declines in adolescent pregnancy in the United States: the contribution of abstinence and improved contraceptive use. Am J Public Health. 2007 Jan;97(1):150-6. doi: 10.2105/AJPH.2006.089169. Epub 2006 Nov 30. PMID 17138906
- [Background] Sonfield A, Hasstedt K, Gold RB. Moving Forward: Family Planning in the Era of Health Reform, New York: Guttmacher Institute, 2014. https://www.guttmacher.org/report/moving-forward-family-planning-era-health-reform; accessed March 1, 2018.
- [Background] Frost JJ, Darroch JE, Remez L. Improving contraceptive use in the United States. Issues Brief (Alan Guttmacher Inst). 2008;(1):1-8. PMID 18561392
- [Background] Santelli JS, Morrow B, Anderson JE, Lindberg LD. Contraceptive use and pregnancy risk among U.S. high school students, 1991-2003. Perspect Sex Reprod Health. 2006 Jun;38(2):106-11. doi: 10.1363/psrh.38.106.06. PMID 16772192
- [Background] Fine LC, Mollen CJ. A pilot study to assess candidacy for emergency contraception and interest in sexual health education in a pediatric emergency department population. Pediatr Emerg Care. 2010 Jun;26(6):413-6. doi: 10.1097/PEC.0b013e3181e0578f. PMID 20502389
- [Background] Ziv A, Boulet JR, Slap GB. Emergency department utilization by adolescents in the United States. Pediatrics. 1998 Jun;101(6):987-94. doi: 10.1542/peds.101.6.987. PMID 9606224
- [Background] Chernick L, Kharbanda EO, Santelli J, Dayan P. Identifying adolescent females at high risk of pregnancy in a pediatric emergency department. J Adolesc Health. 2012 Aug;51(2):171-8. doi: 10.1016/j.jadohealth.2011.11.023. Epub 2012 Apr 4. PMID 22824448
- [Background] Miller MK, Pickett M, Leisner K, Sherman AK, Humiston SG. Sexual health behaviors, preferences for care, and use of health services among adolescents in pediatric emergency departments. Pediatr Emerg Care. 2013 Aug;29(8):907-11. doi: 10.1097/PEC.0b013e31829ec244. PMID 23903671
- [Background] Walton MA, Resko S, Whiteside L, Chermack ST, Zimmerman M, Cunningham RM. Sexual risk behaviors among teens at an urban emergency department: relationship with violent behaviors and substance use. J Adolesc Health. 2011 Mar;48(3):303-5. doi: 10.1016/j.jadohealth.2010.07.005. PMID 21338903
- [Background] Jaccard J, Levitz N. Counseling adolescents about contraception: towards the development of an evidence-based protocol for contraceptive counselors. J Adolesc Health. 2013 Apr;52(4 Suppl):S6-13. doi: 10.1016/j.jadohealth.2013.01.018. PMID 23535060
- [Background] Zuckerman B, Nathan S, Mate K. Preventing unintended pregnancy: a pediatric opportunity. Pediatrics. 2014 Feb;133(2):181-3. doi: 10.1542/peds.2013-1147. Epub 2014 Jan 27. No abstract available. PMID 24470643
- [Background] Gordon JA, Billings J, Asplin BR, Rhodes KV. Safety net research in emergency medicine: proceedings of the Academic Emergency Medicine Consensus Conference on "The Unraveling Safety Net". Acad Emerg Med. 2001 Nov;8(11):1024-9. doi: 10.1111/j.1553-2712.2001.tb01110.x. PMID 11691663
- [Background] Bernstein SL, D'Onofrio G. Public health in the emergency department: Academic Emergency Medicine consensus conference executive summary. Acad Emerg Med. 2009 Nov;16(11):1037-9. doi: 10.1111/j.1553-2712.2009.00548.x. No abstract available. PMID 20053218
- [Background] Hallfors DD, Iritani BJ, Miller WC, Bauer DJ. Sexual and drug behavior patterns and HIV and STD racial disparities: the need for new directions. Am J Public Health. 2007 Jan;97(1):125-32. doi: 10.2105/AJPH.2005.075747. Epub 2006 Nov 30. PMID 17138921
- [Background] Miller MK, Randell KA, Barral R, Sherman AK, Miller E. Factors Associated With Interest in Same-Day Contraception Initiation Among Females in the Pediatric Emergency Department. J Adolesc Health. 2016 Feb;58(2):154-9. doi: 10.1016/j.jadohealth.2015.10.016. PMID 26802990
- [Background] Miller MK, Champassak S, Goggin K, Kelly P, Dowd MD, Mollen CJ, et al. A brief intervention to reduce adolescent sexual risk behaviors: feasibility and impact. J Adolescent Health. 2014;54(2S):S11.
- [Background] Mollen CJ, Miller MK, Hayes KL, Wittink MN, Barg FK. Developing emergency department-based education about emergency contraception: adolescent preferences. Acad Emerg Med. 2013 Nov;20(11):1164-70. doi: 10.1111/acem.12243. PMID 24238320
- [Background] Miller MK, Hornberger L, Sherman AK, Dowd MD. Acceptability of sexual health discussion and testing in the pediatric acute care setting. Pediatr Emerg Care. 2013 May;29(5):592-7. doi: 10.1097/PEC.0b013e31828e646f. PMID 23611917
- [Background] Chernick LS, Westhoff C, Ray M, Garcia M, Garth J, Santelli J, Dayan PS. Enhancing referral of sexually active adolescent females from the emergency department to family planning. J Womens Health (Larchmt). 2015 Apr;24(4):324-8. doi: 10.1089/jwh.2014.4994. PMID 25860108
- [Background] Mehta SD, Hall J, Lyss SB, Skolnik PR, Pealer LN, Kharasch S. Adult and pediatric emergency department sexually transmitted disease and HIV screening: programmatic overview and outcomes. Acad Emerg Med. 2007 Mar;14(3):250-8. doi: 10.1197/j.aem.2006.10.106. PMID 17331918
- [Background] Silva A, Glick NR, Lyss SB, Hutchinson AB, Gift TL, Pealer LN, Broussard D, Whitman S. Implementing an HIV and sexually transmitted disease screening program in an emergency department. Ann Emerg Med. 2007 May;49(5):564-72. doi: 10.1016/j.annemergmed.2006.09.028. Epub 2006 Nov 20. PMID 17113684
- [Background] Trent M, Chung SE, Burke M, Walker A, Ellen JM. Results of a randomized controlled trial of a brief behavioral intervention for pelvic inflammatory disease in adolescents. J Pediatr Adolesc Gynecol. 2010 Apr;23(2):96-101. doi: 10.1016/j.jpag.2009.06.005. Epub 2009 Sep 3. PMID 19733100
- [Background] Suffoletto B, Akers A, McGinnis KA, Calabria J, Wiesenfeld HC, Clark DB. A sex risk reduction text-message program for young adult females discharged from the emergency department. J Adolesc Health. 2013 Sep;53(3):387-93. doi: 10.1016/j.jadohealth.2013.04.006. Epub 2013 May 23. PMID 23707402
- [Background] Calderon Y, Cowan E, Nickerson J, Mathew S, Fettig J, Rosenberg M, Brusalis C, Chou K, Leider J, Bauman L. Educational effectiveness of an HIV pretest video for adolescents: a randomized controlled trial. Pediatrics. 2011 May;127(5):911-6. doi: 10.1542/peds.2010-1443. Epub 2011 Apr 11. PMID 21482613
- [Background] Mollen CJ, Miller MK, Hayes KL, Barg FK. Knowledge, attitudes, and beliefs about emergency contraception: a survey of female adolescents seeking care in the emergency department. Pediatr Emerg Care. 2013 Apr;29(4):469-74. doi: 10.1097/PEC.0b013e31828a3249. PMID 23528510
- [Background] Miller MK, Mollen CJ, O'Malley D, Owens RL, Maliszewski GA, Goggin K, Kelly P. Providing adolescent sexual health care in the pediatric emergency department: views of health care providers. Pediatr Emerg Care. 2014 Feb;30(2):84-90. doi: 10.1097/PEC.0000000000000076. PMID 24457494
- [Background] Miller MK, Plantz DM, Dowd MD, Mollen CJ, Reed J, Vaughn L, Gold MA. Pediatric emergency health care providers' knowledge, attitudes, and experiences regarding emergency contraception. Acad Emerg Med. 2011 Jun;18(6):605-12. doi: 10.1111/j.1553-2712.2011.01079.x. PMID 21676058
- [Background] Reed JL, Punches BE, Taylor RG, Macaluso M, Alessandrini EA, Kahn JA. A Qualitative Analysis of Adolescent and Caregiver Acceptability of Universally Offered Gonorrhea and Chlamydia Screening in the Pediatric Emergency Department. Ann Emerg Med. 2017 Dec;70(6):787-796.e2. doi: 10.1016/j.annemergmed.2017.04.017. Epub 2017 May 27. PMID 28559031
- [Background] Goyal MK, Teach SJ, Badolato GM, Trent M, Chamberlain JM. Universal Screening for Sexually Transmitted Infections among Asymptomatic Adolescents in an Urban Emergency Department: High Acceptance but Low Prevalence of Infection. J Pediatr. 2016 Apr;171:128-32. doi: 10.1016/j.jpeds.2016.01.019. Epub 2016 Feb 2. PMID 26846572
- [Background] Chernick LS, Schnall R, Higgins T, Stockwell MS, Castano PM, Santelli J, Dayan PS. Barriers to and enablers of contraceptive use among adolescent females and their interest in an emergency department based intervention. Contraception. 2015 Mar;91(3):217-25. doi: 10.1016/j.contraception.2014.12.003. Epub 2014 Dec 12. PMID 25499588
- [Background] Mollen C, Lavelle J, Hawkins L, Ambrose C, Ruby B. Description of a novel pediatric emergency department-based HIV screening program for adolescents. AIDS Patient Care STDS. 2008 Jun;22(6):505-12. doi: 10.1089/apc.2007.0098. PMID 18462077
- [Background] Cowan E, Leider J, Velastegui L, Wexler J, Velloza J, Calderon Y. A qualitative assessment of emergency department patients' knowledge, beliefs, attitudes, and acceptance toward revised HIV testing strategies. Acad Emerg Med. 2013 Mar;20(3):287-94. doi: 10.1111/acem.12090. PMID 23517261
- [Background] Reed JL, Vaughn LM, Pomerantz WJ. Attitudes and knowledge regarding emergency contraception among emergency department adolescents and providers. Pediatr Emerg Care. 2012 Aug;28(8):775-9. doi: 10.1097/PEC.0b013e3182627d14. PMID 22858752
- [Background] Office of Disease Prevention and Health Promotion. Healthy People 2020. https://www.healthypeople.gov/2020/topics-objectives/topic/family-planning/objectives; Accessed December 12, 2017.
- [Background] National Institutes of Health. NICHD Research Priorities; https://www.nichd.nih.gov/grants-contracts/research-areas/priorities; Accessed January 4, 2018.
- [Background] National Center for Health Statistics. National Survey of Family Growth, 2013-2015. 2016; https://www.cdc.gov/nchs/nsfg/. Accessed January 15, 2018.
- [Background] Hoopes AJ, Benson SK, Howard HB, Morrison DM, Ko LK, Shafii T. Adolescent Perspectives on Patient-Provider Sexual Health Communication: A Qualitative Study. J Prim Care Community Health. 2017 Oct;8(4):332-337. doi: 10.1177/2150131917730210. Epub 2017 Sep 20. PMID 28929860
- [Background] Kumar MM. Long-Acting Reversible Contraceptives for Adolescents: More Complex Than "First-Line". JAMA Pediatr. 2018 Jan 1;172(1):6-7. doi: 10.1001/jamapediatrics.2017.3520. No abstract available. PMID 29159411
- [Background] Ott MA, Sucato GS; Committee on Adolescence. Contraception for adolescents. Pediatrics. 2014 Oct;134(4):e1257-81. doi: 10.1542/peds.2014-2300. PMID 25266435
- [Background] Madden T, Mullersman JL, Omvig KJ, Secura GM, Peipert JF. Structured contraceptive counseling provided by the Contraceptive CHOICE Project. Contraception. 2013 Aug;88(2):243-9. doi: 10.1016/j.contraception.2012.07.015. Epub 2012 Sep 5. PMID 22959396
- [Background] Haynes MC, Ryan N, Saleh M, Winkel AF, Ades V. Contraceptive Knowledge Assessment: validity and reliability of a novel contraceptive research tool. Contraception. 2017 Feb;95(2):190-197. doi: 10.1016/j.contraception.2016.09.002. Epub 2016 Sep 9. PMID 27621043
- [Background] Oregon Health Authority. Oregon reproductive health program 2015 client satisfaction survey report. 2015; https://public.health.oregon.gov/HealthyPeopleFamilies/ReproductiveSexualHealth/Resources/Documents/County_Data_Sheets/2015_CSS_Statewide.pdf. Accessed January 12, 2017.
- [Background] Mollen CJ, Barg FK, Hayes KL, Gotcsik M, Blades NM, Schwarz DF. Assessing attitudes about emergency contraception among urban, minority adolescent girls: an in-depth interview study. Pediatrics. 2008 Aug;122(2):e395-401. doi: 10.1542/peds.2008-0009. PMID 18676526
- [Background] Guest G, Bunce A, Johnson L. How many interviews are enough?: An experiment with data saturation and variability. Field Methods 2006;18:59.
- [Background] Robin L, Dittus P, Whitaker D, Crosby R, Ethier K, Mezoff J, Miller K, Pappas-Deluca K. Behavioral interventions to reduce incidence of HIV, STD, and pregnancy among adolescents: a decade in review. J Adolesc Health. 2004 Jan;34(1):3-26. doi: 10.1016/s1054-139x(03)00244-1. PMID 14706401
- [Background] Kraut-Becher J, Eisenberg M, Voytek C, Brown T, Metzger DS, Aral S. Examining racial disparities in HIV: lessons from sexually transmitted infections research. J Acquir Immune Defic Syndr. 2008 Mar 1;47 Suppl 1:S20-7. doi: 10.1097/QAI.0b013e3181605b95. PMID 18301130
- [Background] Jemmott JB 3rd, Jemmott LS, Fong GT. Abstinence and safer sex HIV risk-reduction interventions for African American adolescents: a randomized controlled trial. JAMA. 1998 May 20;279(19):1529-36. doi: 10.1001/jama.279.19.1529. PMID 9605896
- [Background] Weeks K, Levy SR, Zhu C, et al. Impact of a school-based AIDS prevention program on young adolescents' self-efficacy skills. Health Educ Res 1995;10:329-344.
- [Background] Kirby DB, Laris BA, Rolleri LA. Sex and HIV education programs: their impact on sexual behaviors of young people throughout the world. J Adolesc Health. 2007 Mar;40(3):206-17. doi: 10.1016/j.jadohealth.2006.11.143. PMID 17321420
- [Background] DiClemente RJ, Salazar LF, Crosby RA. A review of STD/HIV preventive interventions for adolescents: sustaining effects using an ecological approach. J Pediatr Psychol. 2007 Sep;32(8):888-906. doi: 10.1093/jpepsy/jsm056. Epub 2007 Aug 27. PMID 17726032
- [Background] Schwartlander B, Stover J, Hallett T, Atun R, Avila C, Gouws E, Bartos M, Ghys PD, Opuni M, Barr D, Alsallaq R, Bollinger L, de Freitas M, Garnett G, Holmes C, Legins K, Pillay Y, Stanciole AE, McClure C, Hirnschall G, Laga M, Padian N; Investment Framework Study Group. Towards an improved investment approach for an effective response to HIV/AIDS. Lancet. 2011 Jun 11;377(9782):2031-41. doi: 10.1016/S0140-6736(11)60702-2. PMID 21641026
- [Background] Levinson RA, Wan CK, Beamer LJ. The contraceptive self-efficacy scale: analysis in four samples. J Youth Adolesc. 1998 Dec;27(6):773-93. doi: 10.1023/a:1022865900546. PMID 12349803

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents and APPs were enrolled from Emergency Departments of two geographically distinct urban pediatric hospitals.
Groups:
- Contraception Counseling in ED: APPs administer contraception counseling to adolescents.
  Adolescents complete survey and follow up data, and APP completes feasibility data.
- APP Contraception Counseling Training: APPs are trained to conduct a brief contraception counseling session with adolescents in the ED.
Period: Overall Study
Arm/Group | Contraception Counseling in ED | APP Contraception Counseling Training
Started | 108 (The first participant was enrolled on November 13th, 2019. All adolescent participants received counseling in the ED by APP participants. (Single intervention among adolescent group completed by APPs)) | 27 (27 APPs were consented to participate and all APPs were consented during their in-person component of the training.)
Completed | 99 (Last participant enrolled 2/17/2021) | 27
Not Completed | 9 | 0
Not completed — Determined to be ineligible or there was no APP to perform the counseling. | 9 | 0

BASELINE CHARACTERISTICS:
Population: 96 participants were assessed at baseline, received the adolescent counseling intervention and completed outcome information. Please note, no baseline measures were collected for the APP participants.
Groups:
- Adolescent Counseling Intervention; APP Contraception Counseling Training: All adolescent participants will receive contraception counseling.
  Contraception Counseling: Each participant will receive a 10 minute confidential contraception counseling session with an Advanced Practice Provider(APP) in the Emergency Department
  Please note, no baseline measures were collected for APP participants.
- Total: Total of all reporting groups
Arm/Group | Adolescent Counseling Intervention | APP Contraception Counseling Training | Total
Number analyzed (Participants) | 96 | 0 | 96
Age, Categorical [Count of Participants; unit: Participants] — Population: Please note, no baseline measures were collected for APP participants.
  Participants
    <=18 years | 96 | 0 | 96
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: Please note, no baseline measures were collected for APP participants.
  years | 16.8 [15 to 18] |  | 16.8 [15 to 18]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Please note, no baseline measures were collected for APP participants.
  Participants
    Female | 96 | 0 | 96
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Please note, no baseline measures were collected for APP participants.
  Participants
    Hispanic or Latino | 16 | 0 | 16
    Not Hispanic or Latino | 79 | 0 | 79
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: Three of participants enrolled initially were not included in study analysis due to enrollment eligibility errors or having not received contraception counseling. Among the 96 participants remaining who completed study measures and were included in analysis, 45 were enrolled at cmh (site 2).
  Please note, no baseline measures were collected for APP participants.
  Participants
    United States | 96 | 0 | 96

OUTCOME MEASURES:

1. Primary Outcome: Intention to Initiate Contraception
Description: Intention to initiate contraception at Emergency Department (ED) or follow-up visit from survey responses
Time Frame: up to 8 weeks
Population: Those who reported "high intention" to initiate contraception
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Counseling Intervention: All participants will receive contraception counseling.
  Contraception Counseling: Each participant will receive a 10 minute confidential contraception counseling session with an Advanced Practice Provider in the Emergency Department
Arm/Group | Adolescent Counseling Intervention
Number analyzed (Participants) | 96
Participants | 59

2. Secondary Outcome: Contraceptive Care Referral Completion
Description: Participants completed a referral visit for any contraception care
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Counseling Intervention: All participants will receive contraception counseling.
  Contraception Counseling: Each participant will receive a 10 minute confidential contraception counseling session with an Advanced Practice Provider in the Emergency Department
Arm/Group | Counseling Intervention
Number analyzed (Participants) | 96
Participants | 35

3. Secondary Outcome: Initiation of Contraception
Description: Participant has started contraception as evidenced by electronic medical record view and follow-up phone calls or surveys
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Counseling Intervention
Number analyzed (Participants) | 96
Participants | 32

4. Other Pre Specified Outcome: Number of Unique Themes Affecting Decision-Making
Description: Semistructured interviews were conducted and analyzed using grounded theory to elucidate the factors that affect decision-making around contraception initiation. Only a subset of enrolled adolescents participated in interviews which were optional (28 participants).
  Factors were based on a theoretical framework called eTPB, the ecologically expanded theory of planned behavior, relying on attitudes, subjective norms, community, health care and perceived behavioral control factors to explain behavior. Interview analysis yielded the following factors: concerns about contraception side effects and safety, previous experiences with contraception, reasons for using contraception, peer, family and partner influence, social media, pregnancy rates, and access to contraception eduction, provider encounters, confidence in contraception decision making and knowledge, and the ED session characteristics; all of the above factors corresponded with a construct from eTPB.
Time Frame: up to 12 weeks
Population: The total number of unique themes for all participants was reported based on qualitative analysis. 28 adolescents participated in interviews out of the total number of adolescents enrolled in the study. This portion of the study was optional.
Measure: Number; unit: themes
Groups:
- Adolescent Interviews: Participants that received contraception counseling with an Advanced Practice Provider in the Emergency Department and consented to and completed a follow-up interview about their contraception decision-making.
Arm/Group | Adolescent Interviews
Number analyzed (Participants) | 28
themes | 6

ADVERSE EVENTS:
Time Frame: Up to eight weeks
Description: Up to eight weeks after the index ED visit participants were contacted by text message to complete a follow-up survey assessing referral completion and contraception initiation.
Arm/Group | Counseling Intervention | APP Contraception Counseling Training
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/27
Other Adverse Events (participants affected / at risk) | 0/99 | 0/27

LIMITATIONS AND CAVEATS:
Coronavirus (COVID) 19 occurred during the study recruitment period and impacted the duration of time needed to reach our recruitment goals, and our ability to reach our initial recruitment goals. The sample size was recalculated to establish a suitable reduced sample size achievable within the confines of the study enrollment period and study budget.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT04120376/Prot_SAP_000.pdf
  • Informed Consent Form: Advanced Practice Providers (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04120376/ICF_001.pdf
  • Informed Consent Form: Patients (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT04120376/ICF_002.pdf